CLINICAL TRIAL: NCT06329635
Title: Trial of Treatment of Vasospasm Associated With Aneurysmal Subarachnoid Hemorrhage With Intrathecal Injection of Nicardipine: a Multi-center, Prospective, Double-blinded, Randomized Controlled Trial
Brief Title: Treatment of Vasospasm of Aneurysmal Subarachnoid Hemorrhage With Intrathecal Nicardipine - FAST-IT Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Zeguang Ren, Principal Investigator, The Affiliated Hospital Of Guizhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023070K
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Vasospasm
Keywords: Aneurysmal Subarachnoid Hemorrhage; Vasospasm; Delayed cerebral ischemia; Nicardipine; Intrathecal injection
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The assigned "intervention" will be performed only by a separate unblinded dedicated physician who signs the confidential agreement. The attending/investigating physician and patient are blinded to the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Treatment Group (Experimental): The participants in the IT treatment group will be treated with intrathecal nicardipine injection through EVD or LP draining catheter.
  Interventions: Drug: Intrathecal Nicardipine
- Control Group (Sham Comparator): The participants of the control group will receive no intrathecal nicardipine injection through EVD or LP draining catheter.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Intrathecal Nicardipine — First, 6 ml of cerebrospinal fluid is withdrawn from the EVD or LD catheter, and then 4 ml (4mg) of nicardipine is injected into the EVD or LD drain tube, followed by 2 ml normal saline solution, and then the EVD or LD tube is clamped for 2 hours, and then kept open as clinically necessary until the next dose (q12h) of medication.
  Other Names: Treatment group
  Arms: Intrathecal Treatment Group
Other: No intervention — A simulated "intrathecal administration" operation is performed by a dedicated physician who is unblinded to the group assignment, the EVD or LD tube is not opened, and no "drug" is given. The simulated administration process needs to be out of the patient's view (if awake patient) and out of the presence of study team personnel.
  Other Names: Blank control group
  Arms: Control Group

SUMMARY:
To investigate whether patients with cerebral vasospasm associated with aneurysmal subarachnoid hemorrhage have a better prognosis with intrathecal nicardipine injection via extraventricular drainage or lumbar drainage.

DETAILED DESCRIPTION:
Objective:

To investigate whether patients with cerebral vasospasm associated with aneurysmal subarachnoid hemorrhage have a better prognosis with intrathecal nicardipine injection via extraventricular drainage or lumbar drainage.

Design:

This study is a multi-center, prospective, double-blinded, randomized controlled trial.

Interventions:

First, 6 ml of cerebrospinal fluid is withdrawn from the EVD or LD catheter, and then 4 ml of nicardipine hydrochloride is injected into the EVD or LD drain tube, followed by 2 ml of 0.9 % sodium chloride solution (NaCl), and then the EVD or LD tube was clamped for 2 hours after the injection was completed, then kept open as clinically necessary until the next dose (twice a day).

ELIGIBILITY:
Inclusion criteria:

1. Age 18-80.
2. Spontaneous SAH confirmed by head CT.
3. Saccular brain aneurysm is identified and treated, either surgically or endovascularly.
4. SAH Fisher grade >1 or modified Fisher grade >0.
5. EVD placed for acute hydrocephalus, or LD placed for draining bloody CSF as deemed necessary by the treating physician.
6. Any clinical scenario leading to the diagnosis of possible vasospasm, which includes:

   1. Mean flow velocity of MCA >120, or Lindegaard Ratio ( LR ) > 3.
   2. Any intracranial artery including MCA, ACA, PCA, and BA, TCD showed an upward trend of mean flow velocity for 2 consecutive days (>25cm/s/day).
   3. Clinical deterioration including mental status change (GCS score decrease > 2) and focal neurological deficit unable to be attributed to other known neurological reasons.
   4. Evidence of vasospasm on CTA or DSA, or ischemic change by CTP, MRI.
7. Within 14 days of onset of SAH.
8. Informed consent obtained from the patient or family member.

Exclusion criteria:

1. Hunt-Hess Grade 5 or WFNS Grade 5 (no clinical improvement after EVD placement for acute hydrocephalus).
2. Bacterial or distal aneurysms without subarachnoid hemorrhage in the basal cisterns.
3. The treating physician determines that the culprit aneurysm has not been fully repaired, with a very high likelihood of rebleeding in the near term.
4. History of head trauma within the past 3 months.
5. Any recent brain disease within 3 months, such as tumors, stroke, epilepsy, vasculitis, arteriovenous malformation, hydrocephalus, etc.
6. History of psychiatric disorders or seizures within 3 months.
7. Severe concurrent medical conditions.
8. Pregnant women or those of childbearing potential with a positive urine or serum β-human chorionic gonadotropin (HCG) test.
9. Lactating women.
10. Life expectancy of less than 1 year prior to aSAH onset.
11. Pre-morbid mRS score >1.
12. Participation in another randomized clinical trial that may confound the evaluation of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Dichotomized Modified Rankin Scale (mRS) 0-2 vs 3-6 | Day 90±30, Day 365±60.
  The percentage of patients with mRS 0-2

SECONDARY OUTCOMES:
Extended Glasgow Outcome Score (GOS-E). | Day 90±30, Day 365±60.
  Minimum score 1 and maximum score 8 with higher number being better outcome
Modified Rankin Scale ordinal shift with mRS 5 and 6 combined | Day 90±30, Day 365±60.
  Shift analysis looks at transitions across different levels of mRS score, shifting from higher score to lower score means favorable outcome
Dichotomized Modified Rankin Scale (mRS) 0-3 vs 4-6 | Day 90±30, Day 365±60.
  The percentage of patients with mRS 0-3
Mini-Mental State Examination (MMSE) score | Day 90±30, Day 365±60.
  Minimum score 0 and maximum score 30 with higher score being better outcome
Change of National Institutes of Health Stroke Scale (NIHSS) score | At discharge
  NIHSS Scores range from 0 - 42 with higher score being worse outcome
Cerebrospinal fluid shunt surgery rate | Day 90±30, Day 365±60.
  The incidence of CSF shunt surgery
Overall mortality rate | Day 90±30, Day 365±60.
  All etiology of mortality
Rate of CSF infection | Day 30±7
  Diagnosed with fever, positive CSF test including culture.
Rate of any type of new intracranial hemorrhage. | Day 90±30, Day 365±60.
  The incidence of CSF shunt surgery
Adverse Event | Baseline, Day 2-21, Day 90±30, Day 365±60.
  From enrollment to the end of the study, any event meeting the definition of adverse event (AE) was defined as an adverse event, and each occurrence was recorded in a separate adverse event table.
Serious Adverse Event | Baseline, Day 2-21, Day 90±30, Day 365±60.
  During the period from enrollment to the end of the study, any event meeting the definition of serious adverse event (SAE) was defined as serious adverse event, and each occurrence was recorded by a separate adverse event table.

CONTACTS AND LOCATIONS:
Overall Officials: Zeguang Ren, Principal Investigator — Affiliated Hospital of Guizhou Medical University
Locations (28):
- China (28):
  - Affiliated First Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tiantan Hospital, Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Ninth People's Hospital, Chongqing, Chongqing Municipality
  - Southern Medical University Zhujiang Hospital, Guangzhou, Guangdong
  - Affiliated South China Hospital of Shenzhen University, Shenzhen, Guangdong
  - Nanning First People's Hospital, Nanning, Guangxi
  - Jinyang Hospital Affiliated to Guizhou Medical University, Guiyang, Guizhou
  - The Second Affiliated Hospital of Guizhou Medical University, Kaili, Guizhou
  - Liupanshui City People's Hospital, Liupanshui, Guizhou
  - People's Hospital of Qiannan Buyi and Miao Autonomous Prefecture, Guizhou Province, Xingyi, Guizhou
  - Qianxinan Prefecture People's Hospital, Xingyi, Guizhou
  - Xingyi City People's Hospital, Xingyi, Guizhou
  - Qianfengdong Prefecture People's Hospital, Kaili, G
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang Central Hospital, Henan Province, Nanyang, Henan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - The First People's Hospital of Zhenjiang City, Jiangsu Province, Zhenjiang, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Jinggangshan University Affiliated Hospital, Ji’an, Jiangxi
  - Taian Central Hospital, Shandong Province, Tai’an, Shandong
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Airport Hospital of Sichuan University, Chengdu, Sichuan
  - Western Medical University Affiliated Hospital, Luzhou, Sichuan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Khindi T, Macdonald RL, Schweizer TA. Cognitive and functional outcome after aneurysmal subarachnoid hemorrhage. Stroke. 2010 Aug;41(8):e519-36. doi: 10.1161/STROKEAHA.110.581975. Epub 2010 Jul 1. PMID 20595669
- [Background] Vergouwen MD; Participants in the International Multi-Disciplinary Consensus Conference on the Critical Care Management of Subarachnoid Hemorrhage. Vasospasm versus delayed cerebral ischemia as an outcome event in clinical trials and observational studies. Neurocrit Care. 2011 Sep;15(2):308-11. doi: 10.1007/s12028-011-9586-8. PMID 21748502
- [Background] Macdonald RL, Hunsche E, Schuler R, Wlodarczyk J, Mayer SA. Quality of life and healthcare resource use associated with angiographic vasospasm after aneurysmal subarachnoid hemorrhage. Stroke. 2012 Apr;43(4):1082-8. doi: 10.1161/STROKEAHA.111.634071. Epub 2012 Feb 9. PMID 22328549
- [Background] Springer MV, Schmidt JM, Wartenberg KE, Frontera JA, Badjatia N, Mayer SA. Predictors of global cognitive impairment 1 year after subarachnoid hemorrhage. Neurosurgery. 2009 Dec;65(6):1043-50; discussion 1050-1. doi: 10.1227/01.NEU.0000359317.15269.20. PMID 19934963
- [Background] Pegoli M, Mandrekar J, Rabinstein AA, Lanzino G. Predictors of excellent functional outcome in aneurysmal subarachnoid hemorrhage. J Neurosurg. 2015 Feb;122(2):414-8. doi: 10.3171/2014.10.JNS14290. Epub 2014 Dec 12. PMID 25495745
- [Background] Frontera JA, Fernandez A, Schmidt JM, Claassen J, Wartenberg KE, Badjatia N, Connolly ES, Mayer SA. Defining vasospasm after subarachnoid hemorrhage: what is the most clinically relevant definition? Stroke. 2009 Jun;40(6):1963-8. doi: 10.1161/STROKEAHA.108.544700. Epub 2009 Apr 9. PMID 19359629
- [Background] Vergouwen MD, Vermeulen M, van Gijn J, Rinkel GJ, Wijdicks EF, Muizelaar JP, Mendelow AD, Juvela S, Yonas H, Terbrugge KG, Macdonald RL, Diringer MN, Broderick JP, Dreier JP, Roos YB. Definition of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage as an outcome event in clinical trials and observational studies: proposal of a multidisciplinary research group. Stroke. 2010 Oct;41(10):2391-5. doi: 10.1161/STROKEAHA.110.589275. Epub 2010 Aug 26. PMID 20798370
- [Background] Grossen AA, Ernst GL, Bauer AM. Update on intrathecal management of cerebral vasospasm: a systematic review and meta-analysis. Neurosurg Focus. 2022 Mar;52(3):E10. doi: 10.3171/2021.12.FOCUS21629. PMID 35231885
- [Background] Fisher CM, Kistler JP, Davis JM. Relation of cerebral vasospasm to subarachnoid hemorrhage visualized by computerized tomographic scanning. Neurosurgery. 1980 Jan;6(1):1-9. doi: 10.1227/00006123-198001000-00001. PMID 7354892
- [Background] Reilly C, Amidei C, Tolentino J, Jahromi BS, Macdonald RL. Clot volume and clearance rate as independent predictors of vasospasm after aneurysmal subarachnoid hemorrhage. J Neurosurg. 2004 Aug;101(2):255-61. doi: 10.3171/jns.2004.101.2.0255. PMID 15309916
- [Background] Vorkapic P, Bevan JA, Bevan RD. Longitudinal in vivo and in vitro time-course study of chronic cerebrovasospasm in the rabbit basilar artery. Neurosurg Rev. 1991;14(3):215-9. doi: 10.1007/BF00310660. PMID 1944936
- [Background] Wartenberg KE, Schmidt JM, Claassen J, Temes RE, Frontera JA, Ostapkovich N, Parra A, Connolly ES, Mayer SA. Impact of medical complications on outcome after subarachnoid hemorrhage. Crit Care Med. 2006 Mar;34(3):617-23; quiz 624. doi: 10.1097/01.ccm.0000201903.46435.35. PMID 16521258
- [Background] Al-Mufti F, Amuluru K, Damodara N, El-Ghanem M, Nuoman R, Kamal N, Al-Marsoummi S, Morris NA, Dangayach NS, Mayer SA. Novel management strategies for medically-refractory vasospasm following aneurysmal subarachnoid hemorrhage. J Neurol Sci. 2018 Jul 15;390:44-51. doi: 10.1016/j.jns.2018.02.039. Epub 2018 Feb 23. PMID 29801906
- [Background] Murayama Y, Malisch T, Guglielmi G, Mawad ME, Vinuela F, Duckwiler GR, Gobin YP, Klucznick RP, Martin NA, Frazee J. Incidence of cerebral vasospasm after endovascular treatment of acutely ruptured aneurysms: report on 69 cases. J Neurosurg. 1997 Dec;87(6):830-5. doi: 10.3171/jns.1997.87.6.0830. PMID 9384391
- [Background] Yalamanchili K, Rosenwasser RH, Thomas JE, Liebman K, McMorrow C, Gannon P. Frequency of cerebral vasospasm in patients treated with endovascular occlusion of intracranial aneurysms. AJNR Am J Neuroradiol. 1998 Mar;19(3):553-8. PMID 9541318
- [Background] Charpentier C, Audibert G, Guillemin F, Civit T, Ducrocq X, Bracard S, Hepner H, Picard L, Laxenaire MC. Multivariate analysis of predictors of cerebral vasospasm occurrence after aneurysmal subarachnoid hemorrhage. Stroke. 1999 Jul;30(7):1402-8. doi: 10.1161/01.str.30.7.1402. PMID 10390314
- [Background] Rumalla K, Lin M, Ding L, Gaddis M, Giannotta SL, Attenello FJ, Mack WJ. Risk Factors for Cerebral Vasospasm in Aneurysmal Subarachnoid Hemorrhage: A Population-Based Study of 8346 Patients. World Neurosurg. 2021 Jan;145:e233-e241. doi: 10.1016/j.wneu.2020.10.008. Epub 2020 Oct 10. PMID 33049382
- [Background] Pelz DM, Lownie SP, Mayich MS, Pandey SK, Sharma M. Interventional Neuroradiology: A Review. Can J Neurol Sci. 2021 Mar;48(2):172-188. doi: 10.1017/cjn.2020.153. Epub 2020 Jul 16. PMID 32669144
- [Background] Foreman B. The Pathophysiology of Delayed Cerebral Ischemia. J Clin Neurophysiol. 2016 Jun;33(3):174-82. doi: 10.1097/WNP.0000000000000273. PMID 27258440
- [Background] Abruzzo T, Moran C, Blackham KA, Eskey CJ, Lev R, Meyers P, Narayanan S, Prestigiacomo CJ. Invasive interventional management of post-hemorrhagic cerebral vasospasm in patients with aneurysmal subarachnoid hemorrhage. J Neurointerv Surg. 2012 May;4(3):169-77. doi: 10.1136/neurintsurg-2011-010248. Epub 2012 Feb 28. PMID 22374130
- [Background] Dorsch N. A clinical review of cerebral vasospasm and delayed ischaemia following aneurysm rupture. Acta Neurochir Suppl. 2011;110(Pt 1):5-6. doi: 10.1007/978-3-7091-0353-1_1. PMID 21116906
- [Background] Dorhout Mees SM, Kerr RS, Rinkel GJ, Algra A, Molyneux AJ. Occurrence and impact of delayed cerebral ischemia after coiling and after clipping in the International Subarachnoid Aneurysm Trial (ISAT). J Neurol. 2012 Apr;259(4):679-83. doi: 10.1007/s00415-011-6243-2. Epub 2011 Sep 24. PMID 21947244
- [Background] Rosengart AJ, Huo JD, Tolentino J, Novakovic RL, Frank JI, Goldenberg FD, Macdonald RL. Outcome in patients with subarachnoid hemorrhage treated with antiepileptic drugs. J Neurosurg. 2007 Aug;107(2):253-60. doi: 10.3171/JNS-07/08/0253. PMID 17695377
- [Background] Macdonald RL, Rosengart A, Huo D, Karrison T. Factors associated with the development of vasospasm after planned surgical treatment of aneurysmal subarachnoid hemorrhage. J Neurosurg. 2003 Oct;99(4):644-52. doi: 10.3171/jns.2003.99.4.0644. PMID 14567598
- [Background] Crowley RW, Medel R, Dumont AS, Ilodigwe D, Kassell NF, Mayer SA, Ruefenacht D, Schmiedek P, Weidauer S, Pasqualin A, Macdonald RL. Angiographic vasospasm is strongly correlated with cerebral infarction after subarachnoid hemorrhage. Stroke. 2011 Apr;42(4):919-23. doi: 10.1161/STROKEAHA.110.597005. Epub 2011 Feb 24. PMID 21350201
- [Background] Suzuki S, Suzuki M, Iwabuchi T, Kamata Y. Role of multiple cerebral microthrombosis in symptomatic cerebral vasospasm: with a case report. Neurosurgery. 1983 Aug;13(2):199-203. doi: 10.1227/00006123-198308000-00018. PMID 6888700
- [Background] Romano JG, Forteza AM, Concha M, Koch S, Heros RC, Morcos JJ, Babikian VL. Detection of microemboli by transcranial Doppler ultrasonography in aneurysmal subarachnoid hemorrhage. Neurosurgery. 2002 May;50(5):1026-30; discussion 1030-1. doi: 10.1097/00006123-200205000-00016. PMID 11950405
- [Background] Romano JG, Rabinstein AA, Arheart KL, Nathan S, Campo-Bustillo I, Koch S, Forteza AM. Microemboli in aneurysmal subarachnoid hemorrhage. J Neuroimaging. 2008 Oct;18(4):396-401. doi: 10.1111/j.1552-6569.2007.00215.x. Epub 2008 May 19. PMID 18494776
- [Background] Etminan N, Vergouwen MD, Ilodigwe D, Macdonald RL. Effect of pharmaceutical treatment on vasospasm, delayed cerebral ischemia, and clinical outcome in patients with aneurysmal subarachnoid hemorrhage: a systematic review and meta-analysis. J Cereb Blood Flow Metab. 2011 Jun;31(6):1443-51. doi: 10.1038/jcbfm.2011.7. Epub 2011 Feb 2. PMID 21285966
- [Background] Macdonald RL. Delayed neurological deterioration after subarachnoid haemorrhage. Nat Rev Neurol. 2014 Jan;10(1):44-58. doi: 10.1038/nrneurol.2013.246. Epub 2013 Dec 10. PMID 24323051
- [Background] Macdonald RL, Cusimano MD, Etminan N, Hanggi D, Hasan D, Ilodigwe D, Jaja B, Lantigua H, Le Roux P, Lo B, Louffat-Olivares A, Mayer S, Molyneux A, Quinn A, Schweizer TA, Schenk T, Spears J, Todd M, Torner J, Vergouwen MD, Wong GK; SAHIT Collaboration. Subarachnoid Hemorrhage International Trialists data repository (SAHIT). World Neurosurg. 2013 Mar-Apr;79(3-4):418-22. doi: 10.1016/j.wneu.2013.01.006. Epub 2013 Jan 4. PMID 23295631
- [Background] Ganesh A, Luengo-Fernandez R, Wharton RM, Rothwell PM; Oxford Vascular Study. Ordinal vs dichotomous analyses of modified Rankin Scale, 5-year outcome, and cost of stroke. Neurology. 2018 Nov 20;91(21):e1951-e1960. doi: 10.1212/WNL.0000000000006554. Epub 2018 Oct 19. PMID 30341155
- [Background] Rosenberg N, Lazzaro MA, Lopes DK, Prabhakaran S. High-dose intra-arterial nicardipine results in hypotension following vasospasm treatment in subarachnoid hemorrhage. Neurocrit Care. 2011 Dec;15(3):400-4. doi: 10.1007/s12028-011-9537-4. PMID 21468780
- [Background] Akbik F, Waddel H, Jaja BNR, Macdonald RL, Moore R, Samuels OB, Sadan O. Nicardipine Prolonged Release Implants for Prevention of Delayed Cerebral Ischemia after Aneurysmal Subarachnoid Hemorrhage: A Meta-Analysis. J Stroke Cerebrovasc Dis. 2021 Oct;30(10):106020. doi: 10.1016/j.jstrokecerebrovasdis.2021.106020. Epub 2021 Aug 5. PMID 34365121
- [Background] Barth M, Capelle HH, Weidauer S, Weiss C, Munch E, Thome C, Luecke T, Schmiedek P, Kasuya H, Vajkoczy P. Effect of nicardipine prolonged-release implants on cerebral vasospasm and clinical outcome after severe aneurysmal subarachnoid hemorrhage: a prospective, randomized, double-blind phase IIa study. Stroke. 2007 Feb;38(2):330-6. doi: 10.1161/01.STR.0000254601.74596.0f. Epub 2006 Dec 21. PMID 17185636
- [Background] Yokoya S, Hino A, Goto Y, Oka H. Complete relief of vasospasm - Effect of nicardipine coating during direct clipping for the patient with symptomatic vasospasm of subarachnoid hemorrhage. Surg Neurol Int. 2020 Nov 18;11:394. doi: 10.25259/SNI_640_2020. eCollection 2020. PMID 33282456
- [Background] Dayyani M, Sadeghirad B, Grotta JC, Zabihyan S, Ahmadvand S, Wang Y, Guyatt GH, Amin-Hanjani S. Prophylactic Therapies for Morbidity and Mortality After Aneurysmal Subarachnoid Hemorrhage: A Systematic Review and Network Meta-Analysis of Randomized Trials. Stroke. 2022 Jun;53(6):1993-2005. doi: 10.1161/STROKEAHA.121.035699. Epub 2022 Mar 31. PMID 35354302
- [Background] Weyer GW, Nolan CP, Macdonald RL. Evidence-based cerebral vasospasm management. Neurosurg Focus. 2006 Sep 15;21(3):E8. doi: 10.3171/foc.2006.21.3.8. PMID 17029347
- [Background] Sadan O, Waddel H, Moore R, Feng C, Mei Y, Pearce D, Kraft J, Pimentel C, Mathew S, Akbik F, Ameli P, Taylor A, Danyluk L, Martin KS, Garner K, Kolenda J, Pujari A, Asbury W, Jaja BNR, Macdonald RL, Cawley CM, Barrow DL, Samuels O. Does intrathecal nicardipine for cerebral vasospasm following subarachnoid hemorrhage correlate with reduced delayed cerebral ischemia? A retrospective propensity score-based analysis. J Neurosurg. 2021 Jun 4;136(1):115-124. doi: 10.3171/2020.12.JNS203673. Print 2022 Jan 1. PMID 34087804